CLINICAL TRIAL: NCT00942708
Title: Safety and Efficacy of Fluoxetine in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 052009-009; UL1RR024982 (NIH)
Record Dates: First submitted 2009-07-19; First posted 2009-07-21 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Fluoxetine; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluoxetine (Other): Fluoxetine will be added starting at 20 mg and titrated as tolerated to 80 mg daily.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Total dose How to take:
  Week 1-2 20 mg daily Week 3-4 40 mg daily Week 5-6 40 mg BID Week 7-12 40mg BID
  Other Names: Total dose How to take:; Week 1-2 20 mg daily; Week 3-4 40 mg daily; Week 5-6 40 mg BID; Week 7-12 40mg BID

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of open-label fluoxetine for three months among patients with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Idiopathic pulmonary arterial hypertension (PAH) is a life-threatening disorder of uncertain cause that leads to progressive right heart failure and death. Average survival has improved from about 2.8 years in the early 1990s to approximately 5-7 years with current treatments, but most patients will still die of their disease. Two classes of oral medications are approved for use in PAH: endothelin-1 antagonists, and phosphodiesterase-5 inhibitors. Both improve walk distance and symptoms in PAH, but most patients still have continued dyspnea, fatigue and significant elevations in pulmonary pressures. Those who remain severely impaired are generally started on a continuous intravenous prostacyclin. For those who are less ill but still symptomatic, few options are available.

Primary endpoint: the primary endpoint will be change in pulmonary vascular resistance (PVR) measured by right heart catheterization after three months of therapy.

Secondary endpoints

* Six minute walk distance
* QIDS-SR depression scale

Safety and tolerability endpoints will include a tabulation of adverse events to include but not limited to:

* Death
* Hospitalization
* Symptomatic hypotension
* Gastrointestinal side effects
* Depression

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure
2. PAH of the following subtypes: idiopathic PAH WHO functional class II-III
3. Catheterization within one week showing mPAP >=25, wedge or LV end diastolic pressure ≤15, and PVR > 4 wood units, and baseline fick cardiac output results available
4. Age 16-75
5. Able to complete a six minute walk distance
6. Women of childbearing potential*: negative serum pre-treatment pregnancy test + consistently and correctly uses a reliable method of contraception** Oral approved PAH therapy for >3 months with no change in dose for > 1 month

Exclusion Criteria:

1. PAH with connective tissue disease, congenital heart disease, portal hypertension, glycogen storage disease, Gaucher's disease, hereditary hemorrhagic telangiectasia, hemoglobinopathy, myeloproliferative disorders.
2. Moderate to severe obstructive or restrictive lung disease: forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 70% and FEV1 < 60% of predicted value after bronchodilator administration. -or- total lung capacity (TLC) < 60% of predicted.
3. Systemic systolic blood pressure <100 mmHg Breastfeeding
4. Significant liver, renal or other medical disease preventing completion of the study procedures or with life expectancy <12 months, or any other acute or chronic physical impairment (other than dyspnea), limiting the ability to comply with study requirements

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly M Chin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoxetine: In this single arm study, participants begin fluoxetine at 20 mg daily. If tolerated, the dose is increased every 2 weeks as follows:
  Starting dose: 20 mg daily (week 1-2) Next dose: 40 mg daily (week 3-4) Next dose: 40 mg twice daily (week 5-12)
  If unable to tolerate uptitration, participants may remain at a lower dose.
Period: Overall Study
Arm/Group | Fluoxetine
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Fluoxetine: Fluoxetine will be added starting at 20 mg and titrated as tolerated to 80 mg daily.
  Fluoxetine: :
  Week 1-2 20 mg daily Week 3-4 40 mg daily Week 5-12 40 mg BID
Arm/Group | Fluoxetine
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Vascular Resistance (PVR) at Three Months
Description: PVR will be measured by right heart catheterization at baseline and 3 months. Change in PVR will be determined by baseline value minus 3 month value.
Time Frame: Change in PVR at 3 mos (Baseline - 3 months)
Measure: Mean (Standard Deviation); unit: Wood units
Groups:
- Fluoxetine: Fluoxetine will be started at 20 mg and increased every 2 weeks as tolerated to 80 mg daily.
  Week 1-2 20 mg daily Week 3-4 40 mg daily Week 5-12 40 mg twice daily
Arm/Group | Fluoxetine
Number analyzed (Participants) | 5
Wood units | -0.49 (0.49)
Statistical Analysis 1: Comparison: Fluoxetine; Test type: Other — Single group evaluation of change in PVR between 12 weeks and baseline (T-test for one group, 2-sided, p<0.05 considered significant); p = 0.09, t-test, 1 sided

2. Secondary Outcome: Change Between Baseline and Three Month in the QIDS-SR Depression Scale
Description: The Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR) depression scale is a questionnaire completed by the patient. Lower scores are better. Scoring can be interpreted as 7 or less: normal, 8-12: mild depression, 13-16 moderate depression, 17-20 moderate to severe depression and >20 severe depression. Results here show the median change between baseline and 3 months, making a positive change in score indicative of improvement. Total minimum score is 0 and the maximum is 27.
Time Frame: Baseline - 3 months (median change)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 5
units on a scale | 1 [-1 to 10]

3. Secondary Outcome: Change in Six Minute Walk Distance at 3 Months
Description: Six minute walk distance will be measured at baseline and after 3 months of fluoxetine. Change in walk distance (mean and SD) will be reported by taking subtracting baseline values from result at 3 months.
Time Frame: 3 months
Population: All patients completing the 12 week study were analyzed
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Fluoxetine
Number analyzed (Participants) | 5
meters | 10 (48)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Fluoxetine: Fluoxetine will be added starting at 20 mg and titrated as tolerated to 80 mg daily.
  Fluoxetine:
  Week 1-2 20 mg daily Week 3-4 40 mg daily Week 5-12 40mg BID
Arm/Group | Fluoxetine
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=6)
Chest pain or tightness (Cardiac disorders) | 1 (1) — Developed chest pain during a line malfunction event (see other AE). Required hospital admission
Line malfunction (Product Issues) | 1 (6) — Patient was receiving a continuous iv medication (not a study medication) and developed a line problem. Required hospital admission and line replacement.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=6)
Cold (Infections and infestations) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Heartburn (Gastrointestinal disorders) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Lightheadedness (Cardiac disorders) | 1 (1)
Shaking (Nervous system disorders) | 1 (1)
Yawning (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Lack of concentration (Nervous system disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Reflux (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No